CLINICAL TRIAL: NCT03158519
Title: iMETX (Individualized Metabolic RX): a Pilot Study of an Environmental Intervention to Increase Energy Expenditure Among Breast Cancer Survivors
Brief Title: iMETX (Individualized Metabolic RX): a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Kathy Miller, Professor of Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0590
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Physical activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iMETX intervention (Experimental): Individualized exercise recommendation
  Interventions: Behavioral: iMETX intervention

INTERVENTIONS:
Behavioral: iMETX intervention — Pre-intervention the participants will wear the running watch for 3 weeks so that researchers can collect data about their daily routines regarding where and how much energy they expend.
  During the intervention participants will wear the running watch for 12 weeks. Every 1-3 days the participants will be given an individualized recommendation for how to increase their activity via the iMETX application. Participants will be able to provide feedback to the researchers throughout intervention period regarding what works and does not in terms of the recommendations for increasing activity.
  Post-intervention the participants will wear the running watch for 12 weeks so that researchers can collect data in order to determine whether physical activity changes made during the intervention are sustained.

SUMMARY:
The purpose of this study is to test the mechanics and feasibility of delivering an individualized intervention to increase physical activity in breast cancer survivors.

In this study, researchers will test an intervention that uses a commonly worn activity monitor (i.e., global positioning system [GPS] enabled running watch) to see if they can "prescribe" specific ways to increase physical activity that are individually tailored to each participant. The goal is to help participants increase their daily physical activity without having to join a gym or other traditional fitness program. Researchers want to see if they can make specific recommendations (using an application that can be added to a cell phone, tablet and/or computer) on ways participants can slowly increase their activity based upon where they live and work and in a way that is tailored individually to them. For example, participants may be given a route to walk on their lunch break, or new place to park to allow for a longer walk to their job. The goal is to meet participants where they are in their current level of fitness, and to help them think of new and creative ways of increasing activity without the frustration of soreness or risk of injury. As they move more, the recommendations will increase with them.

DETAILED DESCRIPTION:
Objectives The investigators hypothesize that developing an individualized and dynamic exercise intervention (iMETX) that accounts for factors of the built environment will be feasible for breast cancer patients following primary treatment. This pilot study will assess the feasibility and provide preliminary estimates of effectiveness of the environmental intervention for increasing the energy expenditure and energetic capacity of breast cancer patients. The investigators will also explore patient feedback with this intervention and changes in levels of fatigue and quality of life. Experience and data from this initial pilot study will be used to refine the intervention and design subsequent studies to test its effectiveness.

Primary objective Evaluate the feasibility of an individualized, dynamic, environmental physical activity intervention for early stage breast cancer patients following primary treatment.

Secondary objectives

1. Determine a preliminary estimate of effect size of the environmental intervention on energetic capacity (power envelope) as measured by Power Protocol-B
2. Determine a preliminary estimate of effect size of the environmental intervention on average daily EE as measured by a wearable hybrid GPS/accelerometer physical activity monitor
3. Determine the effect of the environment intervention on the physical parameters of BMI and lean body mass
4. Determine the effect of the environmental intervention on patient reported fatigue and quality of life
5. Determine the persistence of changes in average daily EE after the intervention is complete (i.e., when individual movement tasks are no longer suggested).
6. Obtain formal and informal patient feedback throughout and after the intervention to assess satisfaction and perceptions of feasibility
7. Assess safety

Exploratory objectives Blood samples will be collected prior to and following the intervention and banked for future correlative studies, including the following: inflammatory cytokines (high sensitivity C reactive protein and interleukin 6), adipokines (adiponectin and leptin), sex hormones (estradiol, estrone, testosterone, and sex hormone binding globulin), and telomere length. In addition the invstigators will explore correlations of built and social environment characteristics and psychosocial characteristics with pre-intervention and changes in energy expenditure.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years
2. Diagnosis of DCIS or stage I, II, or III breast cancer
3. Completion of all primary therapy (with the exception of ongoing endocrine or trastuzumab therapy), including surgery, radiation, and/or chemotherapy greater than 4 weeks prior to study enrollment
4. Body weight less than 350 lbs., as dictated by the weight limit for DXA scanner
5. Regular access to a smart phone or computer

Exclusion criteria

1. Any condition precluding exercise, including: NYHA class II, III, or IV congestive heart failure, uncontrolled angina, myocardial infarction in the prior 12 months, orthopedic surgery in the previous 6 months or plans for orthopedic surgery during the study period, chronic pulmonary conditions such as uncontrolled asthma (symptoms > 2 days/week) or dyspnea requiring oxygen, symptomatic peripheral vascular disease, symptomatic anemia, uncontrolled psychiatric conditions such as schizophrenia, or any other comorbidity that would interfere with the ability to complete and comply with the study protocol in the opinion of the investigator
2. Locally recurrent or metastatic breast cancer
3. Diagnosis of other active malignancy. Prior treated malignancies in addition to breast cancer are acceptable.
4. Pregnancy
5. Requirement of assistive devices (e.g., cane) for ambulation
6. Plans for moving to a new home or workplace during, pre-, or post-intervention period
7. Elective surgery anticipated during, pre-, or post-intervention period (e.g., breast reconstruction)
8. Inability to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | 24 months
  Percent of enrolled patients who complete study through end of intervention period (week 4-week 15)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Spring Mill Medical Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballinger TJ, Althouse SK, Olsen TP, Miller KD, Sledge JS. A Personalized, Dynamic Physical Activity Intervention Is Feasible and Improves Energetic Capacity, Energy Expenditure, and Quality of Life in Breast Cancer Survivors. Front Oncol. 2021 Apr 12;11:626180. doi: 10.3389/fonc.2021.626180. eCollection 2021. PMID 33912450